# INFORMED CONSENT DOCUMENT FOR THE PATIENT CENTRAL HOSPITAL "DR. IGNACIO MORONES PRIETO" CENTRAL HOSPITAL NEUROLOGY DEPARTMENT

ID:74-19 NCT04698525

Study Protocol document date: February 15, 2019; Statistical Analysis Plan document date: October 20, 2020; Informed Consent Form document date: February 5, 2019.

## **ADULT PATIENT**

| TITLE OF THE DEAD | A DOLL BROTOGOL |
|---|---|
| TITLE OF THE RESEARCH PROTOCOL | |
| "Efficacy of memantine compared with sodium valproate in the prophylactic treatment of | |
| migraine". The randomized controlled clinical trial" | |
| REGISTRATION NUMBER OF THE | ETHICS COMMITTEE PERIOD OF |
| PROTOCOL AUTHORIZED BY THE | EXECUTION OF THE AUTHORIZED |
| RESEARCH | PROTOCOL |
| | / |
| PRINCIPAL INVESTIGATOR AND PERSON | ASSIGNMENT OF THE PRINCIPAL |
| IN CHARGE AT THE HOSPITAL | INVESTIGATOR |
| | Department of Neurology |
| | Internal Medicine Division |
| Dr. Ildefonso Rodríguez Leyva | Dr. Ignacio Morones Prieto" Central |
| | Hospital |
| | Autonomous University of San Luis Potosí |
| | Professional license 763163 |
| CO-INVESTIGATOR | CO-INVESTIGATOR ASSIGNMENT |
| Dra. Damaris Daniela Vazquez Guevara | Neurology Department |
| | Internal Medicine Division |
| | Dr. Ignacio Morones Prieto" Central |
| | Hospital |
| | Autonomous University of San Luis Potosí |
| | Professional license 10045226 |
| DATE OF PRESENTATION OF | 1 |

| DATE OF PRESENTATION OF INFORMED CONSENT |
|------------------------------------------|
| PATIENT IDENTIFICATION NUMBER |

The Neurology Department of the Central Hospital, Dr Ignacio Morones Prieto, is conducting a research study to compare the efficacy of Memantine versus sodium

valproate in the prophylactic treatment of Migraine. This study will include 40 patients for three months, each participant, from July 08 to October 30. It will be conducted in the Outpatient Referral, Emergency Outpatient and Neurology services of the Central Hospital "Dr Ignacio Morones Prieto".

## Information for the patient

Migraine is a neurological disease characterized by headaches with variable duration, usually located in the middle of the head. However, it can also be found in the forehead or the whole head. Most patients report that the pain is throbbing (like a heartbeat) and often accompanied by nausea, vomiting, discomfort, intolerance to light and noise. Some patients are warned of Migraine before the headache with particular symptoms such as blurred vision, flashes of light or stars, tunnel vision, known as aura.

To know if your headache is a Migraine, you should be evaluated by a doctor, because migraine headaches are very intense, Migraine becomes incapacitating causing missed work, school or not being able to perform activities of daily living, is one of the reasons why you should go to a neurologist who will make the diagnosis and assess whether you are a candidate for treatment. The treatment of Migraine is divided into two types: acute, which is given at the time of the migraine attack, and prophylactic, which is given to prevent new migraine attacks and reduce their intensity. The complication of Migraine is that it becomes a chronic disease, which implies migraine attacks more than 15 days a month.

You have been invited to participate in this study because you have been diagnosed with Migraine and are candidates for prophylactic treatment. In this research study, we will compare the efficacy of two types of treatment, one known as sodium valproate, already known as a treatment for Migraine and another that could be a new treatment for Migraine, which is Memantine.

To realize this research, the participants who can be included will be separated into two randomized groups, and each group will have 20 participants. One group will receive sodium Valproate, and the other will receive Memantine. However, neither you nor the physician must know which pharmacological treatment you will be receiving for three months.

## Procedures the patient will undergo

Your participation in this research study is entirely voluntary. If you agree to participate, we will ask you to read this informed consent document carefully and to ask all the necessary questions to the responsible research physician, Dr Ildefonso Rodriguez Leyva, so that he can resolve your doubts. When you no longer doubt what will be done in this study, we will ask you to sign your acceptance to participate at the end of this document. We will also ask you to provide us with general information such as your name, age, weight, height, and medical history; in an interview of approximately 45 minutes, Dr Damaris Daniela Vazquez Guevara will conduct the outpatient area of this hospital. So it will not be necessary to review your clinical record. At the end of this first medical assessment, you will be given a migraine diary to record your migraine attacks and their

characteristics. To keep your data anonymous, you will be assigned a code by which only the research physicians participating in this study will be able to know your identity.

Medical evaluations will be performed every four weeks on five occasions at the Neurology outpatient clinic of the Central Hospital by Dr Damaris Daniela Vazquez Guevara. From the second visit, she will be asked again about the frequency of migraine attacks, if she tolerates the medication and possible adverse effects. In addition, at visits 2, 3, and 4, the research team will provide you with the drug at no cost randomly assigned for four weeks, and at each visit, you will be given a new migraine diary which will be collected at the next visit. At all visits, you will be given a survey to assess the intensity of your migraine attack pain. While you are receiving the drugs, you will be monitored by the team for possible adverse effects.

Dr Vazquez has explained to you in detail what your disease consists of and the importance of having a prophylactic treatment with the goal of decreasing the frequency of your migraine attacks.

## **Benefits to the patient:**

You may benefit by having a favourable response to treatment and decreasing the frequency of migraine attacks. However, you will be collaborating with the research area of the Neurology Department of the Central Hospital, "Dr Ignacio Morones Prieto", and we will not know which medication you will be receiving. This study is intended to evaluate a new prophylactic treatment for Migraine that seems to be well tolerated by patients.

### Benefits to society:

This research study will help to evaluate a new drug for the prophylactic treatment of Migraine. Although there are already have medications indicated for Migraine sometimes, patients do not tolerate it or have no response, which is why this new drug is proposed.

#### Potential risks for the patient:

The potential risks involved in your participation are minimal as it is an interventional study. However, you may experience side effects from the drugs such as nausea, vomiting, weight gain, tremor, hair loss.

However, in the remote case that you feel any other discomfort generated by the research drug, it is necessary to notify Dr Damaris Daniela Vazquez Guevara immediately. She will provide the necessary care, which will not create any cost to you.

You should know that if you present a side effect or adverse reaction to the medications and require hospitalization or treatment, the principal investigator will cover the expenses.

We must comment that you will not receive any payment for participating in the study. However, you will be given a copy of this informed consent document signed by the responsible investigators.

#### **Confidentiality:**

The personal and medical information obtained from you in this study is confidential and will be used only by the research team of this project to analyze and complement the results obtained and will not be available for any other purpose. This information will be combined with that of other participants to carry out the present study. To maintain anonymity, you will be assigned a code for the use of your data.

If you so choose, the investigators responsible for this study may inform your treating physician that you have agreed to participate in this study so that the information obtained may be included in your medical record. For this purpose, we will ask you to indicate whether or not you agree to the above at the end of this document.

The results of this study may be published for scientific purposes in special journals directed to medical personnel, nurses, chemists and researchers related to the health area to make them aware of the possibility of a new prophylactic treatment for Migraine. The results of this study may also be presented at scientific meetings where new findings obtained from this and other studies related to the health and treatment of patients with the same diagnosis are discussed. The clinical data of all participants will be presented anonymously and in such a way that you or any of the patients participating in this study cannot be identified.

According to the General Law of Protection of Personal Data in Possession of Obligated Subjects and the Law of Protection of Personal Data of the State of San Luis Potosi, your data may not be processed, transferred or used for purposes not expressly described in this document. For this reason, it is strictly necessary for the exercise and fulfilment of the powers and obligations expressly provided in the rules governing the actions of the researchers responsible for the study. Furthermore, it complies with a legal mandate; it is necessary for public safety, public order, public health or safeguarding the rights of third parties.

For the use of your data or analysis or handling of your samples and results of the studies described in this document must be informed and requested with due justification to the Research Ethics Committee. This entity will determine the pertinence of the request and, if applicable, authorize a different use for your data, samples and products derived from your models and results. All processes will comply with national and international legislative guidelines and norms and benefit and protect the integrity of the participating actors.

There are Mexican institutions or organizations such as the Ministry of Health, the Federal Commission for the Protection against Health Risks (COFEPRIS), the National Bioethics Commission (CONBIOETICA) or even the Research Ethics Committee (CEI) of this hospital, which are responsible for monitoring the proper handling of personal and medical data. Therefore, you and other patients have been authorized to be used in the conduct of research studies such as this one. Furthermore, these institutions or organizations may request from the researchers to review the procedures that are performed with your information and results. For example, those to verify that correct and ethical use of them; may have access to this information that has been previously

assigned with an identification code when is required.

Participation or withdrawal:

Your participation in this study is voluntary. However, you have been invited to participate due to the characteristics of your disease, to be a candidate to receive prophylactic treatment for Migraine.

You are free to refuse to participate in this research study, but if you decide to join at any time and without explanation, you may revoke or cancel the consent you now sign. Your decision whether or not to participate will in no way affect the medical treatment you receive at the institution for your illness. Suppose you decide to terminate your participation in this study. In that case, you must communicate it to Dr Damaris Daniela Vazquez Guevara. She will provide you with a straightforward document (format) in which you will put some of your data and indicate that you no longer wish to participate in the study. Again, your decision to participate or not will not affect in any way the medical treatment you receive in the institution for your disease.

You will be given a copy of this informed consent form which includes the contact information of the person responsible for this study and the Research Ethics Committee of this hospital to clarify any doubts that may arise.

#### **Ethical Considerations:**

This study is considered higher than minimal risk as it is an interventional study. In addition, you will be randomized between 2 interventions because the investigators responsible for this study will be making decisions regarding your treatment for three months.

We will not ask for your authorization to review your clinical record. Instead, we will only ask you some questions, as we have explained previously.

You will be given a copy of this informed consent, signed by the responsible investigator, including their contact information and the contact information of the Research Ethics Committee of this hospital to clarify any doubts that may arise.

Commitment to answer questions and doubts:

To ask any question, doubt or clarification about this the study of the Double-Blind Randomized Clinical Trial to compare the efficacy of Memantine against Sodium Valproate in the prophylactic treatment of Migraine, or about any adverse reaction related to the medication that you are taking as treatment and that has been indicated by your treating physician, and you can contact:

Dr. Ildefonso Rodriguez Leyva
Department of Neurology
Central Hospital "Dr. Ignacio Morones Prieto".

Av. Venustiano Carranza 2395, Col. Zona Universitaria, San Luis Potosí, S.L.P., C.P. 78290, Tel. 6643759438

Dr. Damaris Daniela Vazquez Guevara

Neurology Department

Central Hospital "Dr. Ignacio Morones Prieto".

Av. Venustiano Carranza 2395, Col. Zona Universitaria, San Luis Potosí, S.L.P., C.P. 78290, Tel. 6643759438

If you have any questions regarding your rights as a participant in the research study, you may also contact a person not involved with the research team of this study:

Dr Emmanuel Rivera Lopez

President of the Research Ethics Committee

Central Hospital "Dr. Ignacio Morones Prieto", Venustiano Carranza Ave.

Venustiano Carranza Av. 2395,

Col. Zona Universitaria, San Luis Potosí, S.L.P., C.P. 78290,

Tel (52-444) 8 34 27 01, Ext. 1710

## **Acceptance of the Informed Consent Document**

If you wish to participate in this research voluntarily, please provide your name, signature and date of this document in the spaces provided below. Your signature means that you agree to the following:

- 1. I have been given complete and adequate information verbally and in writing about the purpose of the study, have had it explained to me that the risks are more significant than minimal because it is an intervention study and the benefits of participating in clear language.
- 2. I have been informed that I may withdraw my consent and terminate my participation in this study at any time without affecting my right to medical care.
- 3. It is my responsibility to ask questions to clarify any points I do not understand regarding my participation in this study. I have asked all questions of the person conducting the consent process and have received satisfactory answers.
- 4. I have not concealed or misrepresented any current medical condition or medical history related to my health. I have answered all questions regarding my health accurately and truthfully.
- 5. I am of legal age and legally capable of giving this consent.
- 6. I agree to participate in this study voluntarily without being pressured or coerced. I understand that my refusal to participate or discontinuation of participation at any time will not result in penalty or loss of benefits to which I am otherwise entitled.

- 7. I understand and agree that the information obtained from the present study may be used to publish these results for academic purposes as part of scientific dissemination and in support of clinical practice. But that at all times, and we will be assigned code that will be used to maintain my anonymity and the confidentiality of my data.
- 8. It has been explained to me that the personal and clinical information that I have consented to provide will preserve my privacy and will be used only for purposes arising from this study.
- 9. The investigators participating in this project have agreed to provide me with updated information obtained during the study when I request it and give me a copy of this informed consent document.
- I, at this moment, agree to participate in the medical study entitled "Efficacy of memantine compared to sodium valproate in the prophylactic treatment of migraine". A randomized controlled clinical trial on a free and voluntary basis.

You are asked to indicate your agreement or disagreement so that the investigators

#### Authorization for the use of clinical data

the above and as explained to me.

responsible for this project can use the clinical data anonymously to realize this research protocol. All the objectives and procedures have been explained to you, and that you have freely and voluntarily provided the; mark with an X your answer: Yes, I give my authorization to the investigators participating in this project to use the clinical data that I have provided to them in the research that they have explained to me. I do not give my permission to the investigators participating in this project to use the clinical data that I have provided to them in the research that they have explained to me. Authorization to inform my treating physician of my participation in this research study and include my results in my clinical record. You are requested to indicate your agreement or disagreement with the investigators responsible for this research study to inform your treating physician. that you have agreed participate in this study with the registration number before the IRB of this hospital and for the results obtained from the measurements of blood flow in the arteries of your brain, which you have consented to be performed, to be included in your clinical record so that they can be used as a reference for your treatment by your treating physician. Please mark your answer with an X: Yes, I give my authorization to the investigators to inform my treating physician of my participation in this research study and to have my results included in my file, following

| I, at this moment, give my permission to the physician of my participation in this research stude following the above and as explained to me. | |
|---|---|
| I, at this moment, agree to participate in the memantine compared to sodium valproate in the randomized controlled clinical trial in a free and vo | prophylactic treatment of migraine". A |
| PATIENT'S NAME | PATIENT'S SIGNATURE OF ACCEPTANCE |
| | ACCEPTANCE |
| DATE INFORMED CONSENT OBTAINED | |
| NAME OF LEGAL REPRESENTATIVE (if necessary) | SIGNATURE OF ACCEPTANCE OF LEGAL REPRESENTATIVE |
| DATE INFORMED CONSENT WAS OBTAINED | RELATIONSHIP |
| ADDRESS / CONTACT PH | HONE NUMBER |
| NAME OF WITNESS 1 | SIGNATURE OF WITNESS 1 |
| DATE | RELATIONSHIP |
| ADDRESS / CONTACT PHONE N | UMBER OF WITNESS 1 |
| NAME OF WITNESS 2 | SIGNATURE OF WITNESS 2 |
| DATE | RELATIONSHIP |
| ADDRESS / CONTACT TELEPHONE | NUMBED OF WITNESS 2 |
| ADDRESS / CONTACT TELEPHONE | NOWDER OF WITNESS 2 |

Dr. Damaris Daniela Vazquez Guevara
(name and signature of the person obtaining the
informed consent)
INVESTIGATOR PARTICIPATING IN THE
PROTOCOL

Dr. Ildefonso Rodríguez Leyva

PRINCIPAL INVESTIGATOR AND
RESPONSIBLE
OF THE RESEARCH PROTOCOL
Department of Neurology
Universidad Autonoma de San Luis Potosí
PROFESSIONAL LICENSE 763163

Dra. Damaris Daniela Vazquez Guevara

CO-INVESTIGATOR
Department of Neurology
Universidad Autónoma de San Luis Potosí
CÉDULA PROFESIONAL 10045226